CLINICAL TRIAL: NCT00765115
Title: Assessment of LY450139-Mediated Inhibition of Amyloid Beta Formation Determined by 13C6-Leucine In Healthy Subjects
Brief Title: A Study of Healthy Subjects to Assess the Effect of LY450139 on Amyloid Beta Peptide Production Rate and or Dose Response.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Office, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 9384; H6L-MC-LFAM
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2008-10-02 (Estimated); Status verified 2008-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — N2-((2S)-2-(3,5-difluorophenyl)-2-hydroxyethanoyl)-N1-((7S)-5-methyl-6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-L-alaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 100 mg LY 450139 oral
  Interventions: Drug: LY450139
- 2 (Experimental): 140 mg LY450139 oral
  Interventions: Drug: LY450139
- 3 (Experimental): 280 mg LY450139 oral
  Interventions: Drug: LY450139
- 4 (Experimental): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: LY450139
  Arms: 1; 2; 3
Drug: placebo
  Arms: 4

SUMMARY:
To test that LY450139, a gamma-secretase inhibitor, will reduce the rate of newly synthesize Amyloid Beta by determining the amount of newly synthesized 13C6 leucine-labeled Amyloid Beta in lumbar cerebrospinal fluid from LY450139 treated subjects compared with placebo treated subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers: Men within the ages of 21 and 50

Exclusion Criteria:

* Have serious or unstable medical conditions
* Have a history of serious infections affecting the brain or head trauma resulting in protracted loss of consciousness within the last 5 years or multiple episodes of head trauma
* Have a history of primary or recurrent malignant disease
* Have a recent laboratory result indicating a clinically significant laboratory abnormality as determined by the investigator
* Have a history of chronic alcohol or drug abuse within the past 5 years
* Have a known history of Human immunodeficiency virus (HIV), afebrile seizures, or clinically significant multiple drug allergies
* Are judged clinically by the investigator to be at serious risk for suicide
* Have electrocardiogram abnormalities obtained at visit 1 that in the opinion of the investigator are clinically significant
* Use of prescription or over the counter medications that cannot safely be discontinued within 14 days prior to visit 2
* Have criteria that would preclude a LP such as allergy to all local anesthetics; have a local infection at the site of the LP or have any medical condition requiring treatment with warfarin or heparin.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Are investigator site personnel directly affiliated with this study and or immediate families.
* Are Lilly employees

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To test hypothesis that LY450139, a gamma-secretase inhibitor, will reduce the rate of synthesis of 13C6-leucine-labeled Aβ (newly synthesized) in lumbar cerebrospinal fluid (CSF). | 0-36 hours post dose

SECONDARY OUTCOMES:
To test the hypothesis that LY450139 has an effect on fractional clearance rate of Amyloid Beta assayed from CSF samples in LY450139-treated subjects compared to placebo-treated subjects. | 0-36 hours post dose
To study and evaluate other biomarkers, such as sAPPB and sAPPA that may enable drug effectiveness to be predicted. | 0-36 hours post dose
To measure concentrations of Amyloid Beta(1-40), Amyloid Beta(1-42), and leucine in CSF by mass spectrometry. | 0-36 hours post dose
To explore the relationship between Amyloid Beta plasma decrease and Amyloid Beta synthesis rate as determined by CSF measurements. | 0-36 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigtive sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, St Louis, Missouri, United States

REFERENCES:
- [Derived] Holtta M, Dean RA, Siemers E, Mawuenyega KG, Sigurdson W, May PC, Holtzman DM, Portelius E, Zetterberg H, Bateman RJ, Blennow K, Gobom J. A single dose of the gamma-secretase inhibitor semagacestat alters the cerebrospinal fluid peptidome in humans. Alzheimers Res Ther. 2016 Mar 7;8(1):11. doi: 10.1186/s13195-016-0178-x. PMID 26948580